CLINICAL TRIAL: NCT00675025
Title: An Open-label Study to Evaluate the Safety of Donepezil Hydrochloride((Aricept®) for up to 1 Year in the Treatment of Cognitive Dysfunction Exhibited by Children With Down Syndrome-Follow-up to a 10-Week,Double-Blind,Placebo-Controlled Trial
Brief Title: Evaluating The Safety Of Donepezil Hydrochloride (Aricept) For Up To 1 Year In The Treatment Of The Cognitive Dysfunction Exhibited By Children With Down Syndrome - Follow-Up To A 10-Week, Double-Blind, Placebo-Controlled Trial
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sufficient evidence of efficacy not met. Discontinuation not based on any safety concerns.
Sponsor: Eisai Inc. (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E2020-A001-220; A2501060 (Other: Pfizer)
Record Dates: First submitted 2008-05-07; First posted 2008-05-08 (Estimated); Results first posted 2021-03-29 (Actual); Last update posted 2021-03-29 (Actual); Status verified 2021-03

CONDITIONS: Down Syndrome
MeSH Terms: conditions — Down Syndrome | interventions — Donepezil

ARMS (1):
- Prior Donepezil-DB (Experimental): All participants started with a dose of 2.5 mg/day (2.5 mL/day). Dose escalations occurred in 2.5 mg/day increments every 2 weeks (steady state levels assumed to have been reached) to a maximum dose of 10 mg/day, according to the participant's weight schedule and the Investigator's judgment of safety and tolerability. Re-titration was done to maintain the blinding of the double-blind study (E2020-A001-219). Doses could be decreased due to tolerability and could be increased or decreased to maintain a maximum dose of 0.1 to 0.2 mg/kg/day based on the participant's weight at clinic visits during the study duration.
  Interventions: Drug: Donepezil hydrochloride (Aricept)

INTERVENTIONS:
Drug: Donepezil hydrochloride (Aricept) — Liquid form Aricept - 5 mg/5 mL donepezil hydrochloride.
  Other Names: Aricept

SUMMARY:
The purpose of this study is to determine the safety of donepezil hydrochloride (Aricept) in children with Down syndrome who have finished the preceding 10-week, double-blind study of donepezil hydrochloride. Medical tests for drug safety will be conducted at each clinic visit.

DETAILED DESCRIPTION:
All children in this study will take donepezil hydrochloride once a day, and will come back to the clinic at 8, 24 and 42 weeks after the study has begun. In between these clinic visits, the clinical staff will telephone the child's parent or caregiver to discuss drug safety observations and possible changes in drug dose. At the end of the study (42 weeks), psychological testing will also be given to determine how well the child is functioning.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Down syndrome (established during study E2020-A001-220).
* Completion of study E2020-A001-219 (NCT00570128 [also known as A2501059]) with no ongoing seroius adverse events and no severe drug reactions.

Exclusion Criteria:

* Weight less than 20 kg.
* Clinically significant conditions affecting absorption, distribution or metabolism of the study medication.
* No reliable parent or caregiver, or unwillingness or inability of parent or caregiver to fulfill the requirements of the study.
* Females of childbearing potential who are not practicing an effective means of birth control.

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 117 (Actual)
Dates: Start 2008-04-04 (Actual); Primary Completion 2008-11-13 (Actual); Study Completion 2008-12-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (31):
- United States (31):
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Child Neurology Associates, PC, Little Rock, Arkansas
  - Midwest Children's Health Research Institute, Los Angeles, California
  - Children's Hospital and Research Center at Oakland, Oakland, California
  - University of California, Irvine Medical Center, Orange, California
  - UCSD Pediatric Pharmacology Research Unit, San Diego, California
  - Rocky Mountain Pediatrics, P.C., Lakewood, Colorado
  - Neufeld Medical Group, Inc., Fort Myers, Florida
  - Miami Children's Hospital, Miami, Florida
  - Miami Children's Hospital - Medical Genetics and Neuro-Developmental Center, Miami, Florida
  - Phoenix Children's Hospital, Miami, Florida
  - Clinical Studies Centers, LLC, St. Petersburg, Florida
  - Northwest Clinical Research Center, West Palm Beach, Florida
  - Road Runner Research, Atlanta, Georgia
  - Hurley Medical Center, Flint, Michigan
  - Saint Mary's Health Care, Grand Rapids, Michigan
  - Washington University School of Medicine, Grand Rapids, Michigan
  - Regions Hospital, Saint Paul, Minnesota
  - Northwest Clinical Research Center, St Louis, Missouri
  - Meridien Research, Lincoln, Nebraska
  - Clinical Research Center of New Jersey, Voorhees Township, New Jersey
  - Division of Genetics and Developmental Behavior, Durham, North Carolina
  - Metrohealth Medical Center, Cleveland, Ohio
  - Valko and Associates, Toledo, Ohio
  - Office of Lazlo Mate, Tulsa, Oklahoma
  - Medical Univ of South Carolina, Charleston, South Carolina
  - Vanderbilt Children's Hospital, Nashville, Tennessee
  - Down Syndrome Clinic of Houston, Houston, Texas
  - Alamo City Clinical Research, LLC, San Antonio, Texas
  - Community Research Foundation, San Antonio, Texas
  - Neuropsychiatric Research Center of Southwest Florida, Bellevue, Washington

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was recruited at 24 centers in the United States during the period of 4 Apr 2008 to 15 Dec 2008. All participants who completed the double-blind (DB) placebo-controlled, 10 week study (Study 2020-A001-219 [NCT00570128]) were offered enrollment in this study.
Pre-assignment Details: The Screening and baseline activities for this study took place on the same day as the Week 10 final visit of the double-blind (DB) study (2020-A001-219 [NCT00570128]).
Groups:
- Prior Donepezil-DB: Participants who received donepezil in the double-blind study E2020-A001-219 (NCT00570128) were continued in this open label extension (OLE) study to be treated with donepezil titrated to achieve a final dose of 0.1 - 0.2 milligram per kilogram per day (mg/kg/day) using liquid formulated at 5 mg/5 milliliter (mL) for up to approximately Week 42.
- Prior Placebo-DB: Participants who received matched placebo in the double-blind study E2020-A001-219 (NCT00570128) were continued in this OLE study to be treated with donepezil titrated to achieve a final dose of 0.1 - 0.2 mg/kg/day using liquid formulated at 5 mg/5 mL for up to approximately Week 42.
Period: Overall Study
Arm/Group | Prior Donepezil-DB | Prior Placebo-DB
Started | 54 | 63
Completed | 0 | 0
Not Completed | 54 | 63
Not completed — Study Terminated by Sponsor | 38 | 42
Not completed — Adverse Event | 6 | 11
Not completed — Lost to Follow-up | 6 | 4
Not completed — Withdrawal by Subject | 4 | 6

BASELINE CHARACTERISTICS:
Groups:
- Prior Donepezil-DB: Participants who received donepezil in the double-blind study E2020-A001-219 (NCT00570128) were continued in this OLE study to be treated with donepezil titrated to achieve a final dose of 0.1 - 0.2 mg/kg/day using liquid formulated at 5 mg/5 mL for up to approximately Week 42.
- Total: Total of all reporting groups
Arm/Group | Prior Donepezil-DB | Prior Placebo-DB | Total
Number analyzed (Participants) | 54 | 63 | 117
Age, Continuous [Mean (Standard Deviation); unit: years] | 13.4 (2.4) | 13.2 (2.2) | 13.2 (3.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 34 | 57
  Male | 31 | 29 | 60
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 4 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 3 | 5
  White | 46 | 55 | 101
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 6 | 1 | 7

OUTCOME MEASURES:

1. Primary Outcome: Change From Visit 1 (Baseline) to Visit 4 or Early Termination in the Vineland Adaptive Behavior Scales, 2nd Edition, Parent/Caregiver Rating Form (VABS-II/PCRF) Sum of the 9 Sub-domain V-scores
Description: VABS-II/PCRF assessed participant's adaptive behaviors on 3 domains (each has 3 sub-domains): Communication (receptive, expressive, written), Daily Living Skills (personal, domestic, community), Socialization (interpersonal relationships, play a leisure time, coping skills). Parent/caregiver rated participant's behavior for sub-domains from 0 (never present) to 2 (always present). Raw scores from sub-domains converted into standardized score(V-scale scores) ranged:1-24 for each sub-domain, mean=15,standard deviation(SD)=3,higher scores=higher level of adaptive functioning and were summed to obtain V-scale composite score ranged 9-216, mean=100,SD=15,higher scores=higher level of adaptive functioning, positive change=improvement in adaptive functioning. Composite and individual analyses, both raw and standardized scores, were not performed due to lack of significant differences between donepezil and placebo in parent study.
Time Frame: Visit 1 (baseline); Early Termination Visit (Week 36)
Population: Analyses were performed on the Intent-to-treat population. The VABS-II/PCRF composite score, individual analyses of each of the 3 domains and the 9 sub-domains by both raw and standardized scores were not performed due to a lack of significant differences between donepezil and placebo subgroups; the data are provided as listings.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Prior Donepezil-DB | Prior Placebo-DB
Number analyzed (Participants) | 44 | 45
units on a scale
  Baseline (Week 10 of DB study) | 87.73 (16.58) | 92.02 (17.51)
  Early termination visit | 89.37 (20.9) | 91.25 (18.45)

ADVERSE EVENTS:
Time Frame: Baseline up to early termination visit (Week 36)
Groups:
- Prior Placebo-DB: Participants who received matched placebo in the double-blind study E2020-A001-219 (NCT00570128) were continued in this OLE study to be treated with donepezil titrated to achieve a final dose of 0.1 - 0.2 mg/kg/day using liquid formulated at 5 mg/5 mL up to approximately Week 42.
Arm/Group | Prior Donepezil-DB | Prior Placebo-DB
All-Cause Mortality (participants affected / at risk) | 0/54 | 0/63
Serious Adverse Events (participants affected / at risk) | 0/54 | 0/63
Other Adverse Events (participants affected / at risk) | 37/54 | 48/63
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Prior Donepezil-DB (N=54) | Prior Placebo-DB (N=63)
Ear pain (Ear and labyrinth disorders) | 2 | 1
Abdominal pain, upper (Gastrointestinal disorders) | 5 | 4
Diarrhea (Gastrointestinal disorders) | 8 | 15
Flatulence (Gastrointestinal disorders) | 0 | 2
Frequent bowel movements (Gastrointestinal disorders) | 0 | 2
Nausea (Gastrointestinal disorders) | 2 | 4
Vomiting (Gastrointestinal disorders) | 4 | 4
Fatigue (General disorders) | 1 | 3
Pyrexia (General disorders) | 1 | 3
Ear infection (Infections and infestations) | 1 | 2
Gastroenteritis viral (Infections and infestations) | 0 | 2
Nasopharyngitis (Infections and infestations) | 2 | 0
Pharyngitis, streptococcal (Infections and infestations) | 2 | 0
Sinusitis (Infections and infestations) | 6 | 8
Upper respiratory tract infection (Infections and infestations) | 2 | 7
Headache (Nervous system disorders) | 1 | 4
Somnolence (Nervous system disorders) | 4 | 1
Abnormal behavior (Psychiatric disorders) | 1 | 3
Aggression (Psychiatric disorders) | 0 | 2
Initial insomnia (Psychiatric disorders) | 2 | 0
Irritability (Psychiatric disorders) | 3 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 4
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 4
Oroparyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Furuncle (Skin and subcutaneous tissue disorders) | 2 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 2

LIMITATIONS AND CAVEATS:
This was an open-label trial that was terminated early by the Sponsor.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other